CLINICAL TRIAL: NCT02563925
Title: A Pilot Study of Brain Irradiation and Tremelimumab in Metastatic Breast Cancer
Brief Title: Brain Irradiation and Tremelimumab in Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-038
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Results first posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Breast Cancer
Keywords: Brain Irradiation; Tremelimumab; 15-038
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiosurgery; tremelimumab; durvalumab

ARMS (1):
- Radiation and Tremelimumab (Experimental): Subjects will get either whole brain radiation treatment (WBRT) or stereotactic radiosurgery (SRS), as per standard of care, with tremelimumab administered every 28 days. Patients, for whom concurrent HER2 directed therapy trastuzumab is indicated, as determined by the treating investigator, will be enrolled in a parallel HER2 directed therapy trastuzumab safety cohort. Protocol Expansion: Dose 1 of tremelimumab & durvalumab (75 mg & 1500 mg, respectively) will ideally be administered 2 days prior to initiation of brain radiotherapy (or between 5 days prior & 3 days after initiation of radiotherapy). Subjects will get either WBRT or SRS, depending on the number & size of their brain metastases. Following the 1st dose, tremelimumab & duvralumab will be administered q28 days from the date of 1st tremelimumab & durvalumab administration, plus or minus 1 week, for 4 cycles. After the 4th cycle, durvalumab will be administered alone until progression of disease or unacceptable toxicity.
  Interventions: Radiation: Brain radiotherapy or Stereotactic Radiosurgery; Drug: Tremelimumab; Drug: HER2 directed therapy; Drug: Durvalumab

INTERVENTIONS:
Radiation: Brain radiotherapy or Stereotactic Radiosurgery
Drug: Tremelimumab
Drug: HER2 directed therapy
Drug: Durvalumab

SUMMARY:
The purpose of this study is to see if the combination of tremelimumab and durvalumab with brain radiation therapy can help treat this type of breast cancer that has spread to the brain.

DETAILED DESCRIPTION:
A Simon 2-stage single-arm design (n=17) will be employed to evaluate for preliminary efficacy. A maximum of 17 subjects will be accrued to the efficacy arm. After the first 3 patients are enrolled in the efficacy arm, a 6 week enrollment hold will be conducted in order to ensure safety before additional patients are enrolled. An interim assessment will then occur after the first 9 subjects have enrolled, and the accrual to this arm will proceed only if a pre-specified futility threshold is met. Patients not requiring continuation of HER2 directed therapy, such as trastuzumab, will be enrolled in this arm.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CNS metastases for whom SRS or WBRT is indicated, as determined by radiation oncologist assessment
* Age 18 and older at the time of consent
* Written informed consent and authorization obtained from the subject/HIPAA-appointed legal representative prior to performing any protocol-related procedures including screening evaluations
* ECOG performance of 0-2 with anticipated life expectancy of ≥12 weeks
* Histologically or cytologically confirmed invasive breast cancer that is HER2-positive (3+ by IHC and/or >2.0 by FISH) if concurrent HER2-directed therapy is planned;
* Non-CNS progression of disease as assessed by the investigator/treating physician, for which a change in systemic therapy is planned OR achievement of stable or responsive non-CNS disease for which a holiday from the current systemic therapy is planned, as assessed by the investigator/treating physician.
* Measurable non-CNS disease, defined by RECIST1.1 criteria
* Recovered from all toxicities associated with prior treatment, to acceptable baseline status or grade 1 or less (for lab toxicities see below limits for inclusion,), except for toxicities not considered a safety risk, such as alopecia or vitiligo. Peripheral neuropathy must be grade 2 or less
* Adequate organ and marrow function, as defined below:
* platelets ≥ 75x 103/μL;
* absolute neutrophil count (ANC) ≥ 1,000/μL;
* hemoglobin ≥ 9.0 g/dL;
* total bilirubin ≤1.5 x ULN (upper limit of normal) except subject with documented Gilbert's syndrome (≤5 x ULN) or liver metastasis, who must have a baseline total bilirubin ≤3.0 mg/dL;
* AST and ALT ≤ 3 x ULN, unless associated with hepatobiliary metastases, in that case ≤5 x ULN
* serum creatinine ≤ 2 mg/dL (or glomerular filtration rate ≥ 50 ml/min as determined by the Cockcroft-Gault equation);
* Negative hepatitis B serologic tests. If positive results are not indicative of active or chronic infection, the subjects can enter the study at the investigator's discretion
* Females of childbearing potential who are sexually active with a non-sterilized male partner must use a highly effective method of contraception prior to the first dose of investigational product, and must agree to continue using such precautions for 6 months after the final dose of investigational product; cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. They must also refrain from egg cell donation for 6 months after the final dose of investigational product;
* Females of childbearing potential are defined as those who are not surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause);
* A highly effective method of contraception is defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. The acceptable methods of contraception
* Non-sterilized males who are sexually active with a female partner of childbearing potential must use a highly effective method of contraception from Days 1 through 90 post last dose. In addition, they must refrain from sperm donation for 90 days after the final dose of investigational product
* LVEF ≥50% for patients enrolling in the HER2 directed therapy arm
* Willing to attempt a baseline tumor biopsy procedure

Exclusion Criteria:

* CNS complications for whom urgent neurosurgical intervention is indicated (e.g., resection, shunt placement)
* Known leptomeningeal metastases not amenable to radiotherapy. Patients receiving radiotherapy for leptomeningeal metastases are eligible
* Received any prior monoclonal antibody against CTLA-4, programmed cell death 1 (PD1) or programmed cell death 1 ligand 1 (PD-L1)
* Subjects with a history of hypersensitivity to compounds of similar biologic composition to tremelimumab or any constituent of the product
* Subjects with a history of hypersensitivity to compounds of similar biologic composition to durvalumab or any constituent of the product;
* Patients unable to obtain MRI for any reason (e.g., due to pacemaker, ferromagnetic implants, claustrophobia, extreme obesity)
* Concurrent enrollment in another therapeutic clinical study or receipt of an investigational product within the last 4 weeks (participation in the survival follow-up period of a study is not an exclusion criterion)
* Medical conditions (aside from newly-diagnosed brain metastases) for which the chronic use of corticosteroids or other immunosuppressive medications are indicated. Note: inhaled and topical steroids are permitted
* Use of immunosuppressive medications within 14 days before the first dose of study drug. The following are exceptions to this criterion: Intranasal, inhaled, topical steroids, or local steroid injections (e.g. intra articular injection); systemic corticosteroids at physiological doses not to exceed 10mg/day of prednisone or its equivalent; steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication).
* Subjects should not be vaccinated with live attenuated vaccines within one month prior to starting tremelimumab treatment
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results
* Any serious uncontrolled medical disorder or active infection that would impair the subject's ability to receive investigational product, such as conditions associated with frequent diarrhea
* Active or history of autoimmune or inflammatory disorders, including inflammatory bowel disease (e.g., colitis, Crohn's), diverticulitis (with the exception of diverticulosis), irritable bowel disease, celiac disease or other serious gastrointestinal chronic conditions associated with diarrhea. Active or history of systemic lupus erythematosus or Wegener's granulomatosis, Sarcoidosis syndrome, Addison's disease, multiple sclerosis, Graves' disease, Hashimoto's thyroiditis, rheumatoid arthritis, hypophysitis, uveitis, etc. Patients without active disease in the last 5 years may be included but only after consultation with the study physician. Note: the following are exceptions to this criterion: Vitiligo or alopecia; patients with hypothyroidism (i.e. following Hashimoto syndrome) stable on hormone replacement; any chronic skin condition that does not require systemic therapy; patients with celiac disease controlled by diet alone;
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frederica's Correction;
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, active peptic ulcer disease or gastritis, and active bleeding diatheses;
* Known history of previous clinical diagnosis of tuberculosis;
* History of allogeneic organ transplant;
* History of leptomeningeal carcinomatosis
* No active, second potentially life-threatening cancer. No history of another primary malignancy except for; malignancy treated with curative intent and no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence; adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; adequately treated carcinoma in situ without evidence of disease;
* Pregnant or breast feeding at time of consent
* Any condition that would prohibit the understanding or rendering of information and consent and compliance with the requirements of this protocol
* Known positive for HIV, chronic or active hepatitis B or C
* Patient is unable to receive IV contrast
* Neuroimaging evidence of midline shift
* Major surgical procedure, as defined by the investigator, within 28 days prior to the first dose of IP. Note: Local surgery or isolated lesions for palliative intent is acceptable.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-09-18 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shanu Modi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Page DB, Beal K, Linch SN, Spinelli KJ, Rodine M, Halpenny D, Modi S, Patil S, Young RJ, Kaley T, Merghoub T, Redmond D, Wong P, Barker CA, Diab A, Norton L, McArthur HL. Brain radiotherapy, tremelimumab-mediated CTLA-4-directed blockade +/- trastuzumab in patients with breast cancer brain metastases. NPJ Breast Cancer. 2022 Apr 19;8(1):50. doi: 10.1038/s41523-022-00404-2. PMID 35440655
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation and Tremelimumab: Subjects will get either whole brain radiation treatment (WBRT) or stereotactic radiosurgery (SRS), as per standard of care, with tremelimumab administered every 28 days. Patients, for whom concurrent HER2 directed therapy trastuzumab is indicated, as determined by the treating investigator, will be enrolled in a parallel HER2 directed therapy trastuzumab safety cohort.
Period: Overall Study
Arm/Group | Radiation and Tremelimumab
Started | 28
Completed | 26
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Radiation and Tremelimumab
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 50 [31 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (irPFS)
Description: will be defined as the time from the first dose of tremelimumab until death or progressive disease, as measured by irRC. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 12 week
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation and Tremelimumab
Number analyzed (Participants) | 28
Participants
  Progressive Disease | 21
  Death | 1
  Stable Disease | 3
  Partial Response | 1
  Not Evaluable | 2

2. Secondary Outcome: Participants Assessed for Toxicity Using the NCI CTCAE 4.0
Description: safety profile assessed with regular physical examination and toxicity assessment using the NCI CTCAE 4.0. Subjects will be followed with regular radiation oncology assessments as per the standard of care.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Radiation and Tremelimumab: Subjects will get either whole brain radiation treatment (WBRT) or stereotactic radiosurgery (SRS), as per standard of care, with tremelimumab administered every 28 days. Patients, for whom concurrent HER2 directed therapy trastuzumab is indicated, as determined by the treating investigator, will be enrolled in a parallel HER2 directed therapy trastuzumab safety cohort. Protocol Expansion: Dose 1 of tremelimumab & durvalumab (75 mg & 1500 mg, respectively) will ideally be administered 2 days prior to initiation of brain radiotherapy (or between 5 days prior & 3 days after initiation of radiotherapy). Subjects will get either WBRT or SRS, depending on the number & size of their brain metastases. Following the 1st dose, tremelimumab & duvralumab will be administered q28 days from the date of 1st tremelimumab & durvalumab administration, plus or minus 1 week, for 4 cycles. After the 4th cycle, durvalumab will be administered alone until progression of disease or unacceptable toxicity.
  Brain radiotherapy or Stereotactic Radiosurgery
  Tremelimumab
  HER2 directed therapy
  Durvalumab
Arm/Group | Radiation and Tremelimumab
Number analyzed (Participants) | 28
Participants | 28

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Radiation and Tremelimumab
All-Cause Mortality (participants affected / at risk) | 27/28
Serious Adverse Events (participants affected / at risk) | 20/28
Other Adverse Events (participants affected / at risk) | 26/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation and Tremelimumab (N=28)
Abdominal Distension (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 3
Alanine aminotransferase increased (Investigations) | 1
Ascites (Gastrointestinal disorders) | 2
Aspartate aminotransferase increased (Investigations) | 2
Ataxia (Nervous system disorders) | 1
Blood bilirubin increased (Investigations) | 1
Breast pain (Reproductive system and breast disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Colitis (Gastrointestinal disorders) | 3
Confusion (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Death NOS (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 2
Dysphasia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Esophagitis (Gastrointestinal disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Neck edema (General disorders) | 1
Neoplasms ben/mal/unk (inc cyst/polyp) Other, spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Neutrophil count decreased (Investigations) | 1
Pain (General disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Platelet count decreased (Investigations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Somnolence (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation and Tremelimumab (N=28)
Anorexia (Metabolism and nutrition disorders) | 14
Nausea (Gastrointestinal disorders) | 11
Fatigue (General disorders) | 10
Weight loss (Investigations) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 9
Colitis (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 5
Headache (Nervous system disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Dizziness (Nervous system disorders) | 4
Dry Mouth (Gastrointestinal disorders) | 4
Dysgeusia (Nervous system disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Alkaline phosphatase increased (Investigations) | 3
Ataxia (Nervous system disorders) | 3
Pain (General disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3
Alanine aminotransferase increased (Investigations) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anemia (Blood and lymphatic system disorders) | 2
Aspartate aminotransferase increased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gen disorders & admin site conditions Other, spec (General disorders) | 2
Hypothyroidism (Endocrine disorders) | 2
Investigations - Other, specify (Investigations) | 2
Malaise (General disorders) | 2
Resp, thoracic & mediastinal disorder Other, spec (Respiratory, thoracic and mediastinal disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-29): https://cdn.clinicaltrials.gov/large-docs/25/NCT02563925/Prot_SAP_000.pdf